CLINICAL TRIAL: NCT02828319
Title: Clinical Study of Z-213 in Subjects With Iron-deficiency Anemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zeria Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Z213-03
Record Dates: First submitted 2016-06-23; First posted 2016-07-11 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Iron Deficiency Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency

ARMS (1):
- Z-213 (Experimental)
  Interventions: Drug: Z-213

INTERVENTIONS:
Drug: Z-213 — The total iron dosage is calculated based on hemoglobin value and the patients' weight, IV on day 1, 8 and 15 (if needed)

SUMMARY:
To confirm the safety and efficacy of Z-213 until 12 weeks after start of Z-213 administration in patients with iron deficiency Anemia

ELIGIBILITY:
Inclusion Criteria:

* Patients with iron deficiency anemia

Exclusion Criteria:

* Patients with anemia caused by conditions other than iron deficiency
* Patients with abnormal laboratory test values at screening for Serum phosphorus, Aspartate aminotransferase, Alanine aminotransferase
* Patients with liver, kidney or circulatory system disease
* Patients with a history or present illness that is a malignant tumor or autoimmune disease
* Patients who underwent intravenous administration of an iron preparation, administration of an erythropoiesis stimulation agent or blood transfusion within 8 weeks before the screening
* Patients who underwent oral administration of an iron preparation (including an over-the-counter drug or supplement) within 4 weeks before the screening

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-07; Primary Completion 2017-05 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Drug Reactions | 12 weeks
Number of participants with Adverse Events | 12 weeks

SECONDARY OUTCOMES:
Maximum change in Hb value | 12 weeks
Change in Hb value | 12 weeks
Proportion of responders | 12 weeks
Proportion of subjects with normalization in Hb value | 12 weeks
Proportion of cumulative dosage | 12 weeks
Number of doses to total dose achieved | 12 weeks
Time to total dose achieved | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Tokyo, Japan